CLINICAL TRIAL: NCT05476614
Title: Testing the Efficacy of Social Robot-led Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamFace Technologies, LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-001
Record Dates: First submitted 2022-05-15; First posted 2022-07-27 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Testing the Efficacy of Social Robot-led Yoga
Keywords: yoga; mindfulness; robot
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Participants will be grouped at random into social robot-instructed yoga or human-instructed yoga.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social robot-instructed yoga group (Experimental): A socially assistive robot will be programmed to instruct 10-14 yoga postures for a group of 20-25 older adults. The yoga session will also include meditation and centering exercises.
  Interventions: Other: Yoga (Robot-instructed)
- Human-instructed yoga group (Active Comparator): A human yoga instructor will lead 10-14 yoga postures for a group of 20-25 older adults. The yoga session will also include meditation and centering exercises.
  Interventions: Other: Yoga (Human-instructed)

INTERVENTIONS:
Other: Yoga (Robot-instructed) — Yoga that is instructed by a social robot
  Arms: Social robot-instructed yoga group
Other: Yoga (Human-instructed) — Yoga that is instructed by a human
  Arms: Human-instructed yoga group

SUMMARY:
Research demonstrates that yoga is beneficial for the older adults with or nearing mild cognitive impairment. Social robots are increasingly being used as companions and caregivers for older adults with or nearing MCI . The purpose of this study is to test the efficacy of social robot-led yoga for older adults with or nearing MCI. The study hypothesizes that social robot-led yoga is similar in effectiveness to human-led yoga across a range of measures.

DETAILED DESCRIPTION:
Research demonstrates that yoga is beneficial for the older adults with or nearing mild cognitive impairment. Social robots are increasingly being used as companions and caregivers for older adults with or nearing MCI. The purpose of this study is to test the efficacy of social robot-led yoga for older adults with or nearing MCI. The study hypothesizes that social robot-led yoga is similar in effectiveness to human-led yoga across a range of measures.

A group of approximately 40-50 older adults (65+) will follow a yoga routine twice per week for 12 weeks taught by either a social robot or human instructor. Details of the yoga instruction can be found below. Yoga sessions will be conducted at an assisted living facility in Denver, Colorado.

Prior to, at the midway point, and after the yoga intervention, researchers will measure participants for the following:

1. Range of motion, overhead flexion: Ryan, the social robot, can scan participants using infrared cameras and create a digital remembrance of their end range of overhead flexion. n = 40 participants will complete the range of motion assessment prior to intervention, midway through the intervention (week 6), post intervention (week 12), and at follow up (week 18).
2. Single-leg balance: Ryan, the social robot, can measure the duration of participant single-leg balance. participants will be asked to balance on their nondominant leg for up to 60 seconds. n = 40 participants will complete the single-leg balance assessment prior to intervention, midway through the intervention (week 6), post intervention (week 12), and at follow up (week 18).
3. The Saint Louis University Mental Status examination (SLUMS): the SLUMS questionnaire will be administered to measure cognitive performance. n = 40 participants will complete the slums prior to intervention, midway through the intervention (week 6), post intervention (week 12), and at follow up (week 18). If at any point the participant meets the exclusion criteria based on SLUMS score, they will be removed from the study.
4. The patient health questionnaire (PHQ-9): researchers will administer the PHQ-9 to measure depression. n = 40 participants will complete the phq-9 prior to intervention, midway through the intervention (week 6), post intervention (week 12), and at follow up (week 18).
5. Kentucky inventory of mindfulness skills (KIMS): researchers will administer the KIMS to measure mindful attention capacity. n= 40 participants will complete the KIMS prior to intervention, midway through the intervention (week 6), post intervention (week 12), and at follow up (week 18).
6. Task engagement: researchers will administer a task engagement questionnaire to measure engagement in the yoga experience. This modified scale will provide a reliable measure of user engagement with both instructors. n = 40 participants will complete the user engagement questionnaire after each yoga session (week 1-12).

At the end of each yoga session, participants will fill out a brief qualitative questionnaire. the questionnaire will ask the following: 1) Please described your experience. 2) What did your instructor do well, where did they struggle? To increase questionnaire brevity, the task engagement questionnaire and qualitative questionnaire are displayed on the same single page of paper.

After six weeks have passed from the date of the last yoga session, participants will be measured one final time as a form of post-participation follow up. Measures will include range of motion, single-leg balance, SLUMS examination, PHQ-9, and KIMS.

Yoga Instruction: Social robot-led yoga will be instructed by Ryan, the social robot. Ryan will be programmed to instruct 10-14 yoga postures in addition to an opening and closing meditation. Each yoga posture will be selected for appropriateness to the developmental age of participants. Several postures will be seated. Others will be standing. Participants will be given the option to stand if they wish and encouraged to move at their own pace. Each posture focuses on creating requisite strength for older adults and correlates to the study's physical measures of single-leg balance and overhead flexion, range of motion. All postures re-enforce each other. Postures will be randomized to ensure variety and updated periodically throughout the study to ensure proper level of challenge and engagement. Updates may include new postures, new verbal or video-based instruction in conjunction with physical instruction changes. Human-led yoga will follow the same format as the social robot-led yoga sessions. Instruction will be 45-minutes of yoga designed with an integrative focus. Human-led yoga will mirror social robot-led yoga in intent, duration, and posture selection.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older.
* SLUMS score of 20-26 will include persons with moderate cognitive impairment
* SLUMS score of >26 will include persons without moderate cognitive impairment
* Verbal skill to interact
* Available for a period of 12 weeks to participate in yoga
* Ability to stand without supports

Exclusion Criteria:

* Age younger than 65 years
* Aggressive behaviors
* Medical diagnosis of dementia or memory loss
* An inability to balance on a single leg without supports
* Acute physical illness that impairs or precludes physical activity
* SLUMS score equal to or below 20, the cutoff for dementia
* A drop in SLUMS score greater than 3 points from the beginning of the study to the midpoint of the study

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Overhead flexion range of motion | At Week 0
  Participant range of motion while standing, arms raise to maximal overhead flexion position. Increased overhead flexion range of motion indicates improved shoulder mobility.
Overhead flexion range of motion | At Week 6
  Participant range of motion while standing, arms raise to maximal overhead flexion position. Increased overhead flexion range of motion indicates improved shoulder mobility.
Overhead flexion range of motion | At Week 12
  Participant range of motion while standing, arms raise to maximal overhead flexion position. Increased overhead flexion range of motion indicates improved shoulder mobility.
Overhead flexion range of motion | At Week 18
  Participant range of motion while standing, arms raise to maximal overhead flexion position. Increased overhead flexion range of motion indicates improved shoulder mobility.
Single-leg balance hold duration | At Week 0
  Participants will hold a balance position unsupported by their arms for a maximum of 60 seconds. Increased single-leg balance hold duration indicates improved fall resilience.
Single-leg balance hold duration | At Week 6
  Participants will hold a balance position unsupported by their arms for a maximum of 60 seconds. Increased single-leg balance hold duration indicates improved fall resilience.
Single-leg balance hold duration | At Week 12
  Participants will hold a balance position unsupported by their arms for a maximum of 60 seconds. Increased single-leg balance hold duration indicates improved fall resilience.
Single-leg balance hold duration | At Week 18
  Participants will hold a balance position unsupported by their arms for a maximum of 60 seconds. Increased single-leg balance hold duration indicates improved fall resilience.

SECONDARY OUTCOMES:
Kentucky Inventory of Mindfulness Skills (KIMS) | At Week 0
  A questionnaire used to assess a participant's ability interact with their environment mindfully. Scoring takes into consideration four facets of mindfulness (Observation, Description, Acting with Awareness, and Judgement). Observation score range (12-60); Description score range (8-40); Act with Awareness score range (10-50); Judgement (9-45). A higher score within the mindfulness attributes of observation, description and awareness indicates increased mindfulness skills. A lower score within the mindfulness attribute of judgement indicates an improvement.
Kentucky Inventory of Mindfulness Skills (KIMS) | At Week 6
  A questionnaire used to assess a participant's ability interact with their environment mindfully. Scoring takes into consideration four facets of mindfulness (Observation, Description, Acting with Awareness, and Judgement). Observation score range (12-60); Description score range (8-40); Act with Awareness score range (10-50); Judgement (9-45). A higher score within the mindfulness attributes of observation, description and awareness indicates increased mindfulness skills. A lower score within the mindfulness attribute of judgement indicates an improvement.
Kentucky Inventory of Mindfulness Skills (KIMS) | At Week 12
  A questionnaire used to assess a participant's ability interact with their environment mindfully. Scoring takes into consideration four facets of mindfulness (Observation, Description, Acting with Awareness, and Judgement). Observation score range (12-60); Description score range (8-40); Act with Awareness score range (10-50); Judgement (9-45). A higher score within the mindfulness attributes of observation, description and awareness indicates increased mindfulness skills. A lower score within the mindfulness attribute of judgement indicates an improvement.
Kentucky Inventory of Mindfulness Skills (KIMS) | At Week 18
  A questionnaire used to assess a participant's ability interact with their environment mindfully. Scoring takes into consideration four facets of mindfulness (Observation, Description, Acting with Awareness, and Judgement). Observation score range (12-60); Description score range (8-40); Act with Awareness score range (10-50); Judgement (9-45). A higher score within the mindfulness attributes of observation, description and awareness indicates increased mindfulness skills. A lower score within the mindfulness attribute of judgement indicates an improvement.
The Patient Health Questionnaire (PHQ-9) | At Week 0
  Depression Questionnaire. Scale minimum value: 0. Scale maximum value: 27). A lower score indicates minimal depression or decreasing depression severity.
The Patient Health Questionnaire (PHQ-9) | At Week 6
  Depression Questionnaire. Scale minimum value: 0. Scale maximum value: 27). A lower score indicates minimal depression or decreasing depression severity.
The Patient Health Questionnaire (PHQ-9) | At Week 12
  Depression Questionnaire. Scale minimum value: 0. Scale maximum value: 27). A lower score indicates minimal depression or decreasing depression severity.
The Patient Health Questionnaire (PHQ-9) | At Week 18
  Depression Questionnaire. Scale minimum value: 0. Scale maximum value: 27). A lower score indicates minimal depression or decreasing depression severity.
The Saint Louis University Mental Status Examination | At Week 0
  A measure of cognitive impairment. Scale minimum value: 0. Scale maximum value: 30. For those with a high school education or greater a score of 27-30 indicates normal function; 21-26 indicates a mild neurocognitive disorder; 0-20 indicates dementia. For those with less than a high school education a score of 25-30 indicates normal function; 20-24 indicates a mild neurocognitive disorder; 0-19 indicates dementia.
The Saint Louis University Mental Status Examination | At Week 6
  A measure of cognitive impairment. Scale minimum value: 0. Scale maximum value: 30. For those with a high school education or greater a score of 27-30 indicates normal function; 21-26 indicates a mild neurocognitive disorder; 0-20 indicates dementia. For those with less than a high school education a score of 25-30 indicates normal function; 20-24 indicates a mild neurocognitive disorder; 0-19 indicates dementia.q
The Saint Louis University Mental Status Examination | At Week 12
  A measure of cognitive impairment. Scale minimum value: 0. Scale maximum value: 30. For those with a high school education or greater a score of 27-30 indicates normal function; 21-26 indicates a mild neurocognitive disorder; 0-20 indicates dementia. For those with less than a high school education a score of 25-30 indicates normal function; 20-24 indicates a mild neurocognitive disorder; 0-19 indicates dementia.
The Saint Louis University Mental Status Examination | At Week 18
  A measure of cognitive impairment. Scale minimum value: 0. Scale maximum value: 30. For those with a high school education or greater a score of 27-30 indicates normal function; 21-26 indicates a mild neurocognitive disorder; 0-20 indicates dementia. For those with less than a high school education a score of 25-30 indicates normal function; 20-24 indicates a mild neurocognitive disorder; 0-19 indicates dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mapoles, MS, Principal Investigator — University of Denver
Locations (1):
- University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brenes GA, Sohl S, Wells RE, Befus D, Campos CL, Danhauer SC. The Effects of Yoga on Patients with Mild Cognitive Impairment and Dementia: A Scoping Review. Am J Geriatr Psychiatry. 2019 Feb;27(2):188-197. doi: 10.1016/j.jagp.2018.10.013. Epub 2018 Oct 25. PMID 30413292
- [Background] Kachouie, R., Sedighadeli, S., Khosla, R., & Chu, M. T. (2014). Socially assistive robots in elderly care: a mixed-method systematic literature review. International Journal of Human-Computer Interaction, 30(5), 369-393.
- [Background] Fan JT, Chen KM. Using silver yoga exercises to promote physical and mental health of elders with dementia in long-term care facilities. Int Psychogeriatr. 2011 Oct;23(8):1222-30. doi: 10.1017/S1041610211000287. Epub 2011 Mar 9. PMID 21385519